CLINICAL TRIAL: NCT00360308
Title: A Multi-centre, Randomised, Double-blind, Placebo and Entacapone Controlled, Parallel Group Study of the Efficacy, Safety and Tolerability of E2007 in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Brief Title: Efficacy, Safety and Tolerability of E2007 in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to lack of efficacy.
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-G000-309; 2006-002937-20 (EudraCT Number)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): matching E2007 and matching entacapone
  Interventions: Drug: Placebo
- E2007 (Active Comparator): 2 mg once daily in the evening, Weeks 0→2 (2 weeks) and 4 mg once daily in the evening, Weeks 2→18.
  Interventions: Drug: E2007
- Entacapone (Active Comparator): 200 mg with each dose of Levodopa.
  Interventions: Drug: E2007

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: E2007
  Arms: E2007
Drug: E2007
  Arms: Entacapone

SUMMARY:
Randomised, double-blind, double dummy, parallel group design. Following the screening period patients will be randomised at the baseline visit, in a 1:1:1 manner, to one of three treatment arms; 4 mg E2007, 200 mg entacapone (with each dose of levodopa) or placebo. The first 4 weeks of the double blind phase will be used to titrate patients on the E2007 arm from 2 mg up to the maintenance dose of 4 mg. Patients randomised to entacapone or placebo will have dummy up titrations to maintain the blind. Following this titration phase, patients will remain on the maintenance dose for a further 14 weeks.

Patients will have visits at 2, 4, 6, 10, 14 and 18 weeks after baseline. A follow up visit will be performed at Week 22.

A home diary will be completed in which patients rate themselves as either:

1. "OFF"
2. "ON" without dyskinesias
3. "ON" with non-troublesome dyskinesias
4. "ON" with troublesome dyskinesias
5. Asleep

These entries will be completed every 30 minutes during the waking day and will be completed for three consecutive days immediately prior to visits at Baseline, Weeks 6, 10, 18 and 22.

At Baseline (Day 0), week 10 and 18 the Unified Parkinson's Disease Rating Scale (UPDRS - Parts I, II , III and IV) will be performed.

At the end of the treatment period (Week 18), patients will undergo final efficacy and safety assessments and will stop taking the study medication they were receiving. They will be seen 4 weeks later for a follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with idiopathic PD fulfilling the (United Kingdom [UK]) Parkinson's disease Society Brain Bank diagnostic criteria, with a good response to levodopa.
2. Patients must have been diagnosed with idiopathic PD at ≥ 30 years of age. In addition the onset of symptoms associated with Parkinson's disease must have occurred ≥ 30 years of age.
3. Patients must have predictable motor fluctuations of the wearing OFF type with the presence of at least 2 hrs of OFF time during the waking day (excluding the morning OFF time) as evidenced by diary cards completed at screening and confirmed by diary data collected in the 3 day diaries completed before randomisation.
4. Before patients are randomised, they must be able to show that they are able to accurately complete the diary cards. During the diary-training period at Screening Visit 1, there must be diary evidence of at least one transition of OFF to ON or from ON to OFF.
5. Patients must rate between II IV on the Hoehn &Yahr (8) scale when in an OFF state.
6. Patients must be taking optimised levodopa (plus dopamine decarboxylase inhibitors [DDI]) therapy (according to the Investigator's opinion) at least 3 times during the waking day (not including bedtime/night time dose) up to a maximum of 8 doses daily (including bedtime/night time dose).
7. Patients who are treated with DA or MAOB inhibitors or other anti-PD drugs must be on optimised and stable doses for at least 4 weeks prior to the Screening visit and must remain stable throughout the study. Only levodopa dosage can be adjusted downwards in the first 6 weeks of the double blind treatment phase.
8. In the Investigator's opinion, patients must be able to distinguish their own motor states and the absence or presence of troublesome or non-troublesome dyskinesias.
9. In the Investigator's opinion, patients are able to complete the study including the completion of the home diary cards and are capable of giving full written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Women of child bearing potential unless infertile (including surgically sterile) or practicing effective contraception (e.g., abstinence, intrauterine device or barrier method plus hormonal method). These patients must have a negative serum B-human chorionic gonadotrophin (B-HCG) test at the initial screening visit (Visit 1) and a negative urine pregnancy test at the baseline visit (Visit 3). These patients must also be willing to remain on their current form of contraception for the duration of the study. Postmenopausal women may be recruited but must be amenorrhoeic for at least 1 year to be considered of non child bearing potential as determined by the Investigator.
3. Patients with a past or present history of drug or alcohol abuse as per Diagnostic and Statistical Manual of Mental Disorders (4th edition; DSM IV) criteria.
4. Patients with a past (within 1 year) or present history of psychotic symptoms requiring anti psychotic treatment. Patients may be taking anti-depressant medication; however, the dose must be stable for 4 weeks prior to the Screening visit. Use of anti psychotic medication including clozapine and quetiapine is prohibited.
5. Patients with a past (within 1 year) or present history of major depression, suicidal ideation or suicide attempts.
6. Patients with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, gastro-intestinal, haematological, endocrine or metabolic systems that might complicate assessment of the tolerability of the study medication.
7. Patients who have a past or present history of liver impairment, neuroleptic malignant syndrome, non traumatic rhabdomyolysis or pheochromocytoma.
8. Patients with significantly elevated liver enzymes (abnormal bilirubin or serum transaminase levels of more than 1.5 times the upper normal limit).
9. Patients with current or prior treatment (within 4 weeks prior to the Screening visit) with medication known to induce the enzyme CYP3A4.
10. Current or prior treatment (within 4 weeks prior to the Screening visit) with pergolide (only applies to patients entering after April 5, 2007), cabergoline (effective as of the date of the IRB/IEC approval of this amendment), tolcapone, methyldopa, budipine, reserpine, quetiapine or intermittent use of either liquid forms of levodopa or subcutaneous apomorphine.
11. Current treatment with non selective MAOA/B or combination of selective MAOA and selective MAOB inhibitors.
12. Patients with a known hypersensitivity to the active substance or to any of the excipients of entacapone.
13. Patients with previous stereotactic surgery (e.g., pallidotomy) for PD or with planned stereotactic surgery during the study period.
14. Patients receiving or with planned (next 6 months) deep brain stimulation.
15. Patients who have received entacapone previously or are currently using entacapone.
16. Patients who have received an investigational product within 4 weeks prior to the Screening visit or patients who have participated in a previous study with E2007.
17. Patients with clinically significant cognitive impairment (Mini Mental State Examination [MMSE] <24 or fulfilling DSM IV criteria for dementia due to PD).
18. Patients with conditions affecting the peripheral or central sensory system unless related to PD (such as mild sensory or pain syndromes limited to OFF periods) that could interfere with the evaluation of any such symptoms caused by the study drug.
19. Patients with any condition that would make the patient, in the opinion of the Investigator, unsuitable for the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, M.D., Study Director — Eisai Inc.
Locations (1):
- Pavillon Riser- Hopital Purpan, Toulouse, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo identical to perampanel (Weeks 0 to 2 one dose per day, Weeks 2 to 18 two doses per day); as well as a placebo identical to entacapone with each dose of levodopa.
- Entacapone: Placebo identical to perampanel (Weeks 0 to 2 one dose per day, Weeks 2 to 18 two doses per day); as well as one entacapone 200 mg dose with each dose of levodopa.
- Perampanel: Perampanel 2 mg (Weeks 0 to 2 one dose per day, Weeks 2 to 18 two doses per day); as well as a placebo identical to entacapone with each dose of levodopa.
Period: Overall Study
Arm/Group | Placebo | Entacapone | Perampanel
Started | 247 | 234 | 242
Completed | 171 | 155 | 154
Not Completed | 76 | 79 | 88
Not completed — Adverse Event | 15 | 14 | 25
Not completed — Abnormal Laboratory Value(s) | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 2
Not completed — Withdrawal by Subject | 11 | 7 | 14
Not completed — Lack of Efficacy | 3 | 0 | 2
Not completed — Other | 2 | 1 | 1
Not completed — Study termination by sponsor | 43 | 55 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Entacapone | Perampanel | Total
Number analyzed (Participants) | 247 | 234 | 242 | 723
Age, Customized [Number; unit: participants]
  <65 years | 131 | 114 | 123 | 368
  ≥65 years | 116 | 120 | 119 | 355
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population was used. The safety population includes the same number of subjects as the Randomized Population except 1 additional subject in the placebo group who was not randomized, but completed the study.
  Participants
    Female | 98 | 98 | 94 | 290
    Male | 149 | 136 | 148 | 433
Race/Ethnicity, Customized [Number; unit: participants] — Race.
  participants
    White | 191 | 176 | 185 | 552
    Asian | 55 | 57 | 57 | 169
    Other | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Daily OFF Time (Hours) to Week 18 (Including LOCF Data)
Description: Efficacy assessments were recorded by subjects using a home diary card. ON state is when medication is providing benefits to mobility, slowness, and stiffness. OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline and Week 18
Population: The Intent-to-Treat (ITT) Population comprised all randomised patients who took at least one dose of study medication or placebo and who had a valid baseline efficacy measure and at least one post-baseline efficacy measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Entacapone | Perampanel
Number analyzed (Participants) | 228 | 221 | 213
Hours | -0.82 [-1.16 to -0.48] | -1.29 [-1.63 to -0.96] | -0.92 [-1.27 to -0.57]

2. Secondary Outcome: Mean Change From Baseline in UPDRS Part II (ADL) Score in Total Daily OFF Time to Week 18 (Including LOCF Data)
Description: Efficacy assessments were recorded by subjects using a home diary card. Unified Parkinson's Disease (PD) Rating Scale (UPDRS) is a standardized assessment of the symptoms and signs of PD. Part II assesses Activities of Daily Living (ADL) based on 13 items, such as speech, hygiene, and falling. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline and Week 18
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Placebo; Perampanel: The total number of subjects reflects 3 fewer subjects due to inavailability of the data
- Entacapone: The total number of subjects reflects 5 fewer subjects due to inavailability of the data
Arm/Group | Placebo | Entacapone | Perampanel
Number analyzed (Participants) | 215 | 210 | 199
Scores on a scale | -1.42 [-2.04 to -0.80] | -2.50 [-3.11 to -1.90] | -1.06 [-1.70 to -0.42]

3. Secondary Outcome: Mean Change From Baseline in UPDRS Part III (Motor) Score in ON State (Hours) to Week 18 (Including LOCF Data)
Description: Efficacy assessments were recorded by subjects using a home diary card. UPDRS is a standardized assessment of the symptoms and signs of PD. Part III assesses motor activity, based on 14 items, such as gait, facial expression, and rigidity. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. ON state is when medication is providing benefits to stiffness, slowness, and tremor.
Time Frame: Baseline and Week 18
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Placebo: The total number of subjects reflects 1 fewer subject due to inavailability of the data
Arm/Group | Placebo | Entacapone | Perampanel
Number analyzed (Participants) | 217 | 215 | 202
Scores on a scale | -1.20 [-2.12 to -0.29] | -3.08 [-3.97 to -2.19] | -1.67 [-2.61 to -0.73]

4. Secondary Outcome: Mean Change From Baseline in Total Daily ON Time (Without Dyskinesias or With Non-troublesome Dyskinesias) (Hours) to Week 18 (Including LOCF Data)
Description: Efficacy assessments were recorded by subjects using a home diary card. ON state is when medication is providing benefits to stiffness, slowness, and tremor.
Time Frame: Baseline and Week 18
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Entacapone | Perampanel
Number analyzed (Participants) | 228 | 221 | 213
Hours | 0.88 [0.52 to 1.24] | 1.10 [0.74 to 1.46] | 0.47 [0.10 to 0.84]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time that the participant signed the informed consent form until 30 days after study drug discontinuation and through the termination visit, whichever is longer.
Description: All AEs were reported on a case report form (CRF). AEs were recorded on subject diaries and by investigators during clinical visits.
Arm/Group | Placebo | Entacapone | Perampanel
Serious Adverse Events (participants affected / at risk) | 6/247 | 8/234 | 11/242
Other Adverse Events (participants affected / at risk) | 39/247 | 63/234 | 66/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=247) | Entacapone (N=234) | Perampanel (N=242)
Cellulitis (Infections and infestations) | 0 | 1 | 1
Otitis Media (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
On and Off Phenomenon (Nervous system disorders) | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=247) | Entacapone (N=234) | Perampanel (N=242)
Nausea (Gastrointestinal disorders) | 9 | 16 | 9
Dizziness (Nervous system disorders) | 7 | 9 | 21
Dyskinesia (Nervous system disorders) | 8 | 27 | 17
On and Off phenomenon (Nervous system disorders) | 16 | 19 | 19
Somnolence (Nervous system disorders) | 4 | 8 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No